CLINICAL TRIAL: NCT04728074
Title: Effects of Vocational Rehabilitation Group Intervention on Motivation and Occupational Self-Awareness in Individuals With Intellectual Disabilities: A Single-Blind, Randomized Control Study
Brief Title: Effects of Vocational Rehabilitation Group Intervention on Motivation and Occupational Self-Awareness in Individuals With Intellectual Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Biruni University (Other)
Responsible Party: Principal Investigator, Orkun Tahir Aran, PhD., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020/34-18
Record Dates: First submitted 2021-01-22; First posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Intellectual Disability
Keywords: self awareness; occupational therapy; vocational rehabilitation; intellectual disability; motivation
MeSH Terms: conditions — Intellectual Disability | interventions — Rehabilitation, Vocational

STUDY DESIGN:
Intervention Model Description: Single blind, randomized control study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The ENtering Employment and SUstaining Work (ENESUW) program consists of 6 main topics which are; "self-awareness", "occupational self-awareness", "taking responsibility", "teamwork and labor division", "problem identification" and "problem solving". The entire program adopts a very plain and easy to understand method of information transmission in order to facilitate lossless comprehension and strengthen the trust relationship between the therapists and the participants.
  The ENESUW program took 8 weeks in total with twice weekly sessions, making up a total of 16 structured group sessions. The group format enabled the participants to learn through meaningful peer interactions and group activities which were supportive of the main learning goals (i.e. group work, labor division and taking responsibility) of the program. The twice weekly sessions were 45 minutes long in order to keep the participants attentive and active throughout the program.
  Interventions: Other: The Entering Employment and Sustaining Work Program; Other: vocational rehabilitation
- control (Active Comparator): The control group also consisted of individuals with ID. They received face to face, individual vocational based occupational therapy approaches, which were twice a week for 8 weeks (approximately 40-45 minutes)
  Interventions: Other: vocational rehabilitation

INTERVENTIONS:
Other: The Entering Employment and Sustaining Work Program — A structured, motivation and self-awareness based group intervention
  Other Names: Occupational therapy - vocational rehabilitation
  Arms: Intervention
Other: vocational rehabilitation — An individual based, focused on desired job or occupation, face-to-face intervention

SUMMARY:
This study is an intervention study that investigates the effects of a group-based approach to motivation and occupational self-awareness of individuals with intellectual disability (ID).

The intervention method was developed by following the intervention mapping method.

An 8 weeks group intervention (twice a week) was applied to individuals with ID which includes; Introduction to intervention and meeting with other group members self-awareness training occupational self-awareness taking responsibility group work and labor division problem identification problem-solving

The entire program was structured and guided by the prepared manual (available upon request from the authors). The manual was prepared by the authors of this study to ensure consistency between different sessions and groups. All sessions were diffusively explained in the manual as well as the individual session booklets. The supervisors were able to follow the structure of the sessions from those booklets. Additionally, there were visual materials for each session as in; presentations, graphics, and photographs. The program supervisors (therapists) met once every week to discuss the progress, participation, and overall status of each participant.

Homework assignments were utilized to facilitate learning. Families were not included directly in the group sessions, however were informed about the homework assignments. Homework assignments consisted of very basic mental practice and reenactment regarding the session's topic and concepts. Families were also included in the final week's sessions since graduation certificates were handed out during these sessions and also small celebrations were carried out.

ELIGIBILITY:
Inclusion Criteria:

1. being between the ages of 18 and 65,
2. Not being currently working,
3. Having formal intellectual disability diagnosis,
4. Having scored 23 points or less from the Mini Mental State Examination,
5. Being able to understand basic Turkish language and 6) Volunteering to participate in the study

Exclusion Criteria:

1. Having severe communication problems specifically in self-expression,
2. Not being able to continue participating in the study for the projected study duration,
3. Not permitted to participate by legal guardian.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2020-05-12 (Actual)

PRIMARY OUTCOMES:
Occupational Self-Assessment version 2.2 (OSA 2.2) | Change from Baseline and to the 2 months
  Occupational Self-Assessment (OSA) is a comprehensive assessment which was designed to collect information regarding the individuals' occupational self-awareness. The OSA is an entirely self-reported tool regarding occupational competence and value. The 21 item OSA evaluates skills (item 1-11), habituation (12-16) and volition (17-21). Each item contains two sets of 4-point Likert scales, the first scale is about the individuals' performance in various activities (1- I have a lot of problem doing this, 2 - I have some difficult doing this, 3 - I do this well, and 4 points = I do this extremely well) and the second scale is about the values of those activities for the individual 1 - This is not important to me, 2 - This is important to me, 3 -This is more important to me; and 4- This is most important to me)
Objective Achievement Motivation Test - OLMT): | Change from Baseline and to the 2 months
  The OLMT is a test which is used for Job & Career replacement and academic testing by assessing examinee's achievement motivation under different circumstances. The OLMT consists of 3 subtests, these 3 subtests include a particular stimulus that motivates respondent's performance: the task itself, setting own goals, and from competition. The test also evaluates the match or mismatch between the set goals and actual performance (aspiration level). For testing; the respondent requires to move a prescribed route cell by cell by pressing two buttons (red and green) repeatedly in ten seconds. For the aspiration level, the respondent sets a goal for the test and tries to accomplish the set goal by performing the first test. The final part the respondent competes against a virtual opponent whose speed is slightly above the mean of the first two tests of the respondent. The scoring of the test is performed by a special software

CONTACTS AND LOCATIONS:
Overall Officials: Hülya Kayıhan, Prof, Study Chair — Occupational Therapy, head of department
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kocman A, Weber G. Job Satisfaction, Quality of Work Life and Work Motivation in Employees with Intellectual Disability: A Systematic Review. J Appl Res Intellect Disabil. 2018 Jan;31(1):1-22. doi: 10.1111/jar.12319. Epub 2016 Dec 21. PMID 28000421
- [Background] Wehman P, Chan F, Ditchman N, Kang HJ. Effect of supported employment on vocational rehabilitation outcomes of transition-age youth with intellectual and developmental disabilities: a case control study. Intellect Dev Disabil. 2014 Aug;52(4):296-310. doi: 10.1352/1934-9556-52.4.296. PMID 25061773